CLINICAL TRIAL: NCT00506805
Title: A Phase 1, Open-label, Dose-escalation Study Of The Safety And Pharmacokinetics Of SNX-5422 Mesylate In Subjects With Refractory Solid Tumor Malignancies Or Non-Hodgkin's Lymphoma
Brief Title: Safety And Pharmacology Study Of SNX-5422 Mesylate In Subjects With Refractory Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Esanex Inc. (Industry)
Collaborators: Serenex, Inc. (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1311001; SNX-5422-CLN1-001
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Cancer
Keywords: solid tumor malignancy; Hsp90
MeSH Terms: conditions — Neoplasms | interventions — SNX-5422

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: SNX-5422

INTERVENTIONS:
Drug: SNX-5422 — dose escalated, tablets every other day; undetermined duration until disease progression

SUMMARY:
Hsp90 is a chemical in the body that is involved in promotion of cancer. SNX-5422 is an experimental drug that blocks Hsp90. It is being evaluated for safety and efficacy in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* histologically confirmed solid tumor malignancy
* refractory to available therapy or for which no therapy is available
* adequate organ function

Exclusion Criteria:

* CNS malignancy
* significant GI disease
* at risk for prolonged QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
adverse events and other safety assessments | continuous

SECONDARY OUTCOMES:
tumor response measured by X-rays or scans | after every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Nashville, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1311001&StudyName=Safety%20And%20Pharmacology%20Study%20Of%20SNX-5422%20Mesylate%20In%20Subjects%20With%20Refractory%20Solid%20Tumor%20Malignancies